## Pilot study of morphological and functional evaluation of adult flat foot by weight bearing CT and gait analysis before and after corrective surgery

**Sponsor**: Istituto Ortopedico Rizzoli

PI: Dr.ssa Lisa Berti

The adult idiopathic flat foot represents a very frequent condition, which afflicts a high percentage of population with different levels of severity and different clinical and functional consequences. This complex foot deformity includes morphological alterations in 3D: valgus of the hindfoot, flattening of the plantar arch and supination of the forefoot. From the functional point of view, flat foot is a syndrome characterized by multiple static and dynamic deformities with the prevalent pronation of the subtalar joint. This complexity explains difficulties in the evaluation of this syndrome and even today the wide debate on indications for surgical treatment and on morphological and functional outcomes.

Morphological weight bearing CT parameters and functional analysis (using "Gait analysis") can implement the evaluation of the flat foot. Weight bearing CT is useful to verify the severity of the 3D deformities typical of flat foot, while kinematic and kinetic variables of gait is able to quantify the functional improvements of the foot after surgery.

The objective of the study consists in morphological and functional evaluation of the adult idiopathic flat foot with a combination of weight bearing CT and "Gait analysis" before and after corrective surgery (arthrodesis of the subtalar joint according to Grice).

Weight bearing CT parameters: position of the calcaneus in 3D (with respect to talus, tibia, midfoot and forefoot) and medial longitudinal arch of the foot.

Gait Analysis parameters: spatio-temporal parameters, multisegmental kinematics of the ankle-foot complex (in coronal, transverse and sagittal planes), medial longitudinal arch and forces.

Clinical examination parameters: VAS of the foot, Foot Posture Index, Foot function Index.

These assessments are performed in a group of 20 patients recruited consecutively and candidates for surgery to correct the adult flat foot according to the Grice technique.

Evaluations are realized by weight bearing CT and by Gait analysis in the pre-operative phase and at a 6-months follow-up from the intervention.

## References

Mann RA. Acquired flatfoot in adults. ClinOrthopRelat Res. 1983Dec;(181):46-51.

Deland JT. Adult-acquired flatfoot deformity. J Am AcadOrthop Surg. 2008Jul;16(7):399-406. Review.

Mosier-LaClair S, Pomeroy G, Manoli A 2nd. Operative treatment of the difficult stage 2 adult acquired flatfoot deformity. Foot Ankle Clin. 2001Mar;6(1):95-119..

1Francisco R, Chiodo CP, Wilson MG. Management of the rigid adult acquired flatfoot deformity. Foot Ankle Clin. 2007 Jun;12(2):317-27.

1Kelly IP, Easley ME. Treatment of stage 3 adult acquired flatfoot. Foot Ankle Clin. 2001 Mar;6(1):153-66.

- 1 Johnson KA, Strom DE. Tibialis posterior tendon dysfunction. Clin Orthop Relat Res. 1989 Feb;(239):196-206.
- 1 Myerson MS. Adult acquired flatfoot deformity: treatment of dysfunction of the posterior tibial tendon. Instr Course Lect. 1997;46:393-405.
- 1Bluman EM, Title CI, Myerson MS. Posterior tibial tendon rupture: a refined classification system. Foot Ankle Clin. 2007 Jun;12(2):233-49.
- 1 Parsons S, Naim S, Richards PJ, McBride D. Correction and prevention of deformity in type II tibialis posterior dysfunction. Clin Orthop Relat Res. 2010 Apr;468(4):1025-32.
- 1 Grice DS. An extra-articular arthrodesis of the subastragalar joint for correction of paralytic flat feet in children. J Bone Joint Surg Am 1952 46:533-541.
- 1 Bacardi BE, Rubin SZ, Turf RM. Complications of the Grice-Green operation. J Foot Surg 1989; 28:325-332.
- Chigot PL, Sananes P: Grice arthrodesis: new indications and technical variant. Rev Chir Orthop Reparatrice Appar Mot 1965; 51:53-65.
- Seymour N, Evans DK. A modification of the Grice subtalar arthrodesis. J Bone Joint Surg Br. 1968 May;50(2):372-5.
- Mann RA, Beaman DN, Horton GA. Isolated subtalar arthrodesis. Foot Ankle Int. 1998 Aug;19(8):511-9.
- Kadakia AR, Haddad SL. Hindfoot arthrodesis for the adult acquired flat foot. Foot Ankle Clin. 2003 Sep;8(3):569-94
- Mann RA, Beaman DN. Double arthrodesis in the adult. ClinOrthopRelat Res. 1999 Aug;(365):74-80 Fortin PT, Walling AK. Triple arthrodesis. ClinOrthopRelat Res. 1999 Aug;(365):91-9.
- Easley ME, Trnka HJ, Schon LC, Myerson MS.Isolatedsubtalar arthrodesis J Bone Joint Surg Am. 2000 May;82(5):613-24
- Barg A, Bailey T, Richter M, de Cesar Netto C, Lintz F, Burssens A, et al. Weightbearing Computed Tomography of the Foot and Ankle: Emerging Technology Topical Review. Foot & Ankle International. 2018;39(3):376–86.
- Carrino JA, Al Muhit A, Zbijewski W, Thawait GK, Stayman JW, Packard N, et al. Dedicated conebeam CT system for extremity imaging. Radiology. 2014;270(3):816–24.
- Tuominen EKJ, Kankare J, Koskinen SK, Mattila KT. Weight-Bearing CT Imaging of the Lower Extremity. American Journal of Roentgenology 2013;200(1):146–8.
- Colin F, Horn Lang T, Zwicky L, Hintermann B, Knupp M. Subtalar Joint Configuration on Weightbearing CT Scan. Foot & Ankle International 2014;35(10):1057–62.
- Lepojärvi S, Niinimäki J, Pakarinen H, Koskela L, Leskelä H. Rotational Dynamics of the Talus in a Normal Tibiotalar Joint as Shown by Weight-bearing Computed Tomography. The Journal of Bone and Joint Surgery 2016;98(7):568–75.
- Hirschmann A, Pfirmann CWA, Klammer G, Espinosa N, Buck FM. Upright Cone CT of the hindfoot: Comparison of the non-weight-bearing with the upright weight-bearing position. European Radiology 2014;24(3):553–8.
- Burssens A, Peeters J, Buedts K, Victor J, Vandeputte G. Measuring hindfoot alignment in weight bearing CT: A novel clinical relevant measurement method. Foot and Ankle Surgery. 2016;22(4):233–8.
- Cody EA, Williamson ER, Burket JC, Deland JT, Ellis SJ. Correlation of Talar Anatomy and Subtalar Joint Alignment on Weightbearing Computed Tomography With Radiographic Flatfoot Parameters. Foot & Ankle International 2016;37(8):874–81.
- Lintz F, Welck M, Bernasconi A, Thornton J, Cullen NP, Singh D, et al. 3D Biometrics for Hindfoot Alignment Using Weightbearing CT. Foot Ankle Int 2017;38(6):684–9.

Caravaggi P, Lullini G, Berti L, Giannini S, Leardini A. Functional evaluation of bilateral subtalar arthroereisis for the correction of flexible flatfoot in children: 1-year follow-up. Gait Posture. 2018 Jun 11;64:152-158.

Caravaggi P, Lullini G, Leardini A, Berti L, Vannini F, Giannini S. Functional and clinical evaluation at 5-year follow-up of a three-component prosthesis and osteochondral allograft transplantation for total ankle replacement. Clin Biomech (Bristol, Avon). 2015 Jan;30(1):59-65.

Malerba F, Benedetti MG, Usuelli FG, Milani R, Berti L, Champlon C, Leardini A. Functional and clinical assessment of two ankle arthrodesis techniques. J Foot Ankle Surg. 2015 May Jun;54(3):399-405.

Berti L, Vannini F, Lullini G, Caravaggi P, Leardini A, Giannini S. Functional evaluation of patients treated with osteochondral allograft transplantation for post-traumatic ankle arthritis: one year follow-up. Gait Posture. 2013 Sep;38(4):945-50.

Caravaggi P, Benedetti MG, Berti L, Leardini A. Repeatability of a multi-segment foot protocol in adult subjects. Gait Posture. 2011 Jan;33(1):133-5.

Leardini A, Benedetti MG, Berti L, Bettinelli D, Nativo R, Giannini S. Rear-foot, mid-foot and fore-foot motion during the stance phase of gait. Gait Posture. 2007 Mar;25(3):453-62.

Levinger P, Murley GS, Barton CJ, Cotchett MP, McSweeney SR, Menz HB. A comparison of foot kinematics in people with normal- and flat-arched feet using the Oxford Foot Model. Gait Posture. 2010.

Hunt AE, Smith RM. Mechanics and control of the flat versus normal foot during the stance phase of walking. Clin Biomech (Bristol, Avon). 2004 May;19(4):391-7.

Buldt AK, Levinger P, Murley GS, Menz HB, Nester CJ, Landorf KB. Foot posture is associated with kinematics of the foot during gait: A comparison of normal, planus and cavus feet. Gait Posture. 2015 Jun;42(1):42-8.

Buldt AK, Murley GS, Butterworth P, Levinger P, Menz HB, Landorf KB. The relationship between foot posture and lower limb kinematics during walking: A systematic review. Gait Posture. 2013 Jul;38(3):363-72.